CLINICAL TRIAL: NCT05115838
Title: A Phase 2a, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Radiopaque Matrix MK-8591 Implant in Participants at Low-Risk for HIV-1 Infection
Brief Title: Radiopaque Matrix MK-8591 Implant in Participants at Low-Risk for Human Immunodeficiency Virus Type 1 (HIV-1) Infection (MK-8591-043)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 8591-043; MK-8591-043 (Other: Merck); 2021-003414-39 (EudraCT Number)
Record Dates: First submitted 2021-11-02; First posted 2021-11-10 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Human Immunodeficiency Virus; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — islatravir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Islatravir 47 mg (Experimental): Participants receive an ISL 47 mg implant for approximately 52 weeks. A subset of participants will receive a second implant for 12 weeks after removal of the first implant.
  Interventions: Drug: Islatravir
- Islatravir 52 mg (Experimental): Participants receive an ISL 52 mg implant for approximately 52 weeks. A subset of participants will receive a second implant for 12 weeks after removal of the first implant.
  Interventions: Drug: Islatravir
- Islatravir 57 mg (Experimental): Participants receive an ISL 57 mg implant for approximately 52 weeks. A subset of participants will receive a second implant for 12 weeks after removal of the first implant.
  Interventions: Drug: Islatravir
- Placebo (Placebo Comparator): Participants receive a placebo implant for approximately 52 weeks. A subset of participants will receive a second implant for 12 weeks after removal of the first implant.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Islatravir — ISL 47, 52, or 57 mg implantable rod placed subdermally on the upper arm.
  Other Names: MK-8591
  Arms: Islatravir 47 mg; Islatravir 52 mg; Islatravir 57 mg
Drug: Placebo — Placebo implantable rod placed subdermally on the upper arm.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of an islatravir (ISL)-eluting implant. Participants will receive an implant placed in the upper arm for approximately 52 weeks with 8 weeks of follow-up in the Base Study. A subset of participants will also receive a second implant for an additional 12 weeks before 8 weeks of follow-up in the Substudy.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health
* Is confirmed human immunodeficiency virus (HIV)-uninfected
* Is at low risk of HIV infection
* For males, uses contraception in accordance with local regulations regarding contraception use for those participating in clinical trials
* For females, is not pregnant or breastfeeding and one of the following applies:
* Is not a participant of childbearing potential (POCBP)
* Is a POCBP and uses an acceptable contraception method or is abstinent

Exclusion Criteria:

* Has an active diagnosis of hepatitis (B or C) due to any cause
* Has a history of malignancy ≤5 years before signing informed consent
* Has a history or current evidence of any condition that might confound study results or interfere with study participation
* Has a history of keloid in upper arm or presence of tattoo, scar, or other physical finding that could interfere with implant placement (the contralateral arm may be used if the findings are limited to 1 arm)
* Is taking or is expected to take immunosuppressants during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-04 (Estimated); Primary Completion 2025-10-02 (Estimated); Study Completion 2025-10-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with ≥1 adverse events (AEs) | Up to 60 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants withdrawing from study treatment due to adverse event (AE) | Up to 52 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Plasma concentration of islatravir (ISL) 12 weeks after placement of an ISL-eluting implant (ISL C12weeks) | Week 12
  Plasma ISL C12weeks will be determined.
Plasma concentration of islatravir (ISL) 52 weeks after placement of an ISL-eluting implant (ISL C52weeks) | Week 52
  Plasma ISL C52weeks will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com